CLINICAL TRIAL: NCT05128019
Title: Can the Use of the Conversation Tool Individual Challenge Inventory Tool (ICIT) by General Practitioners Increase Coping of the Patients?
Brief Title: Use of the Individual Challenge Inventory Tool (ICIT) by General Practitioners
Acronym: ICIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Erik L Werner, Professor, University of Oslo
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NSD368367
Record Dates: First submitted 2021-10-19; First posted 2021-11-19 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Medical Unexplained Physical Symptoms (MUPS); Subjective Health Complaint
Keywords: MUPS, SHC, sick leave, Communication tool, General practice

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Controlled Trial with an intervention group and a control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 50 GPs will recruit 10 patients each from their daily practice, to take part in the study. They will offer the patients a session of unspecified length or number of consultations, to follow the conversation tool ICIT
  Interventions: Behavioral: ICIT
- Control (No Intervention): 50 GPs will recruit 10 patients each from their daily practice, to take part in the study. They will however, only receive standard routine care and follow-up by their GP.

INTERVENTIONS:
Behavioral: ICIT — Patients in the intervention group will receive a number of consultations with their GP based on the ICIT
  Arms: Intervention

SUMMARY:
Many patients in general practice present symptoms that do not refer to specific pathology. We refer to these patients at Medical Unexplained Physical Symptoms (MUPS). Practice and research have well documented that these patients frustrate most General Practitioners (GPs). They also produce a lot of unnecessary investigations and are overrepresented on sick-listing. The conversational tool Individual Challenge Inventory Tool (ICIT) offers an aid for the GPS to the consultation and aims to increase the patients' coping abilities with their health challenges. The aim of the study is to investigate whether patients experience such increased coping following a session of consultations with their GP based on ICIT.

DETAILED DESCRIPTION:
The study is a Cluster Randomized Controlled Trial (cRCT) with GPs as clusters. We plan to includ 50 GPs to participate as intervention group and 50 GPs as controls. Each cluster will include 10 patients. GPs in the intervention group will be trained in the use of ICIT through a 30 hours course, partly digital and partly in presence. The participants will receive lectures on the background for the conversation tool, and the study, and will practice on each other. At the end of the study, also the 50 GPs of the control group will be invited to an identical course.

The outcome of the study is any changes of the patients coping abilities. If the symptoms cannot be healed, a goal for the patients will be to reduce the impact of the symptoms. In practice, this is to reuptake normal activities, including work, in spite of pain, fatigue or mood disturbances. Through the ICIT, the patients will be challenged to look at themselves in a broader spectrum and decide for themselves which activities are possible to reuptake and making a thorough plan for doing so.

The patients will be treated by their regular GP across several meetings and they will agree on a specific plan across weeks or months to achieve their individual goal.

The patients of the GPs in the control group will represent identical medical symptoms and will be treated and followed by their GP as usual. They will, however, be informed and asked to consign to participate in the study, and will respond to the same questionnaires as the patients in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a condition the GP deems as MUPS (unspecific og generalized pain, fatigue or mood disturbances without being depressed)
* Patients must be deemed satisfactory clinical examined without specific findings
* Patients must be able to speak and understand Norwegian language without interpreter
* Patients must sign on a consignment form

Exclusion Criteria:

* Patients must not have any well defined psychiatric diagnosis
* Patients must not have any alcohol or drug abuse
* Patients must not be using more than 10 mg Benzodiasepine per day

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-05-21 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Patients' assessment of personal quality of life | One year
  Patients Global Impression of Change (PGIC)
Patients' experiences at the encounter | One year
  Mean change on score at the Patient Experiences Questionnaire (PEQ)

SECONDARY OUTCOMES:
The primary outcome is any change in patient's coping strategies | One year
  Mean change on score at the Patient Activation Measure (PAM) in both groups

OTHER OUTCOMES:
Single question | One year
  Patients will be asked about their own anticipation of return to work

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abrahamsen C, Reme SE, Wangen KR, Lindbaek M, Werner EL. The effects of a structured communication tool in patients with medically unexplained physical symptoms: a cluster randomized trial. EClinicalMedicine. 2023 Oct 6;65:102262. doi: 10.1016/j.eclinm.2023.102262. eCollection 2023 Nov. PMID 37855023